CLINICAL TRIAL: NCT06301919
Title: Use of N-Butyl Cyanoacrylate in Transarterial Emergency Embolization : a "Real-life" Retrospective Monocentric Study
Brief Title: Use of N-Butyl Cyanoacrylate in Transarterial Emergency Embolization
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN042024/CHUSTE
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-03

CONDITIONS: Haemostasis Embolisation
Keywords: Emergency; Hemostatic agent; NBCA bleeding; Trans-arterial embolisation
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Included patients: All patients referred to our hospital and treated by TAE with NBCA, based on clinical decisions in emergency and CT scan.
  Interventions: Other: Clinical data; Other: Imaging data; Other: Biological data

INTERVENTIONS:
Other: Clinical data — Collecting data from the medical record.
Other: Imaging data — Collecting data from the medical record.
Other: Biological data — Collecting data from the medical record.

SUMMARY:
NBCA is a synthetic biodegradable cyanoacrylate basis glue, modified by the addition of a monomer with adhesive, hemostatic, and antiseptic properties.

Its use requires a steep learning curve to control emulsification of the NBCA/lipiodol mixture, and injection, to avoid non-target embolization.

The aim of this retrospective monocentric study was to evaluate safety and efficacy of use of NBCA as embolic agent in emergency setting.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to our hospital and treated by TAE with NBCA, based on clinical decisions in emergency and CT scan.

Exclusion Criteria:

* Patients lost for follow-up, patients without preoperative CT.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated by TAE with NBCA, based on clinical decisions in emergency and CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of technical success | Month : 1
  Analysis of angiographic results.

SECONDARY OUTCOMES:
Assessment of clinical success | Month : 1
  Disappearance of signs and symptoms of bleeding during the 30 days of follow-up after WT
Assessment of clinical success | Month : 1
  No endoscopic treatment
Assessment of clinical success | Month : 1
  No surgical intervention
Assessment of clinical success | Month : 1
  No repeat WT
Assessment of clinical success | Month : 1
  Absence of death due to massive blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Rémi GRANGE, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No